CLINICAL TRIAL: NCT07100184
Title: Efficacy and Safety of Disitamab Vedotin in Combination With Radiotherapy for Patients With HER2-Expressing High-Risk or Very High-Risk Non-Muscle Invasive Bladder Cancer
Brief Title: RC48 in Combination With Radiotherapy for HER2-Expressing NMIBC Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-RT-01
Record Dates: First submitted 2025-07-21; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-06

CONDITIONS: HER2-expressing High-risk or Very High-risk NMIBC Without Visible Foci of Disease After TURBT
Keywords: non-muscle invasive bladder cancer; NMIBC; HER-2; Disitamab Vedotin; Radiotherapy
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Arm (Experimental): patients with HER2-expressing high-risk or very high-risk non-muscle invasive bladder cancer (NMIBC) without visible foci of disease after transurethral resection of bladder tumor (TURBT)
  Interventions: Drug: Disitamab Vedotin combined with Radiotherapy

INTERVENTIONS:
Drug: Disitamab Vedotin combined with Radiotherapy — Disitamab Vedotin (RC-48) injection 2mg/kg, Q2w for 4 circles before radiotherapy and 2mg/kg, Q3w for 8 circles after radiotherapy; Radiotherapy (Whole bladder dose: 25 Gy in 5 doses, QD)

SUMMARY:
This study is an open, single-arm, single-center exploratory clinical study to explore the efficacy and safety of Disitamab Vedotin (RC-48) in combination with radiotherapy for the treatment of patients with HER2-expressing high-risk or very high-risk non-muscle invasive bladder cancer (NMIBC) without visible foci of disease after transurethral resection of bladder tumor (TURBT). The study plans to enroll 30 patients with high or very high risk HER2-expression NMIBC without visible lesions after TURBT. The study includes a screening period, a treatment period, and a survival follow-up period. This is a single-center study conducted at the Peking University First Hospital, and the PI is Prof. CuiJian Zhang.

ELIGIBILITY:
Inclusion Criteria:

1. voluntarily agree to participate in the study and sign an informed consent form;
2. male or female, age ≥18 years;
3. disease fulfillment:

   1. the patient's disease status was determined by at least two associate or chief physicians to be free of visible lesions to the naked eye after transurethral bladder tumor electrodessication;
   2. A definitive postoperative pathologic diagnosis of non-muscle invasive bladder cancer with >50% of its major tissue component being uroepithelial carcinoma (migratory cell carcinoma);
   3. Completion of TURBT within 4 weeks prior to study administration and completion of immediate chemotherapy infusion (chemotherapy agent is mitomycin);
   4. Absence of focal lymph node metastasis as well as distant metastasis confirmed by imaging (including but not limited to thoracoabdominopelvic CT/MR or PET/CT) within 6 weeks prior to enrollment, i.e., N0M0;
   5. Subject's NMIBC risk grouping is consistent with a high or very high risk group:
4. patient refuses or is unfit to receive BCG infusion; BCG intolerance or progression of BCG therapy;
5. the subject meets 2+ or 3+ HER2 expression by immunohistochemistry (IHC) of tumor tissue obtained by TURBT within 4 weeks;
6. a score of 0-1 on the ECOG Physical Status Scale;
7. adequate cardiac, bone marrow, hepatic, and renal functions

Exclusion Criteria:

1. combined extravesical (i.e., urethral, ureteral, or renal pelvic) uroepithelial cancer;
2. have received any other antineoplastic therapy, such as chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc., within 4 weeks prior to study dosing, excluding 1 instillation of chemotherapy completed immediately after TURBT;
3. has not recovered to CECAT 5.0 grade 0-1 from an adverse event caused by a previously applied antineoplastic agent within 2 weeks prior to initiation of study drug administration;
4. who have had major surgery within 4 weeks prior to the start of study dosing or are scheduled to have major surgery during the study period;
5. Serum virology: a) Positive HBsAg with a positive HBVDNA copy number. b) Positive HCVAb with a positive HBVDNA copy number. c) Positive HBsAg with a positive HBVDNA copy number. d) Positive HBsAg with a positive HBV DNA copy number;
6. have received a live vaccine within 4 weeks prior to the start of study drug administration or plan to receive any vaccine during the study period;
7. heart failure classified by the New York Heart Association (NYHA) as Grade 3 or higher;
8. a serious arterial/venous thrombotic event or cardiovascular accident such as deep vein thrombosis, pulmonary embolism, cerebral infarction, cerebral hemorrhage, myocardial infarction, etc., except for lacunar cerebral infarcts, which are asymptomatic and do not require clinical intervention, within the 6 months prior to study dosing;
9. the presence of an active infection requiring systemic therapy, such as active tuberculosis;
10. the presence of systemic diseases or serious comorbidities that, in the judgment of the investigator, are active and not under stable control, including diabetes mellitus, hypertension, cirrhosis of the liver, interstitial pneumonitis, obstructive lung disease, and that would allow subjects to develop complications as a result of receiving intravesical therapy and/or general anesthesia
11. the presence of any other disease, metabolic abnormality, physical examination abnormality, or laboratory test abnormality that, in the judgment of the investigator, gives reason to suspect that the patient has a disease or condition that is unsuitable for the use of the study medication, or that will interfere with the interpretation of the results of the study, or that places the patient at a high risk of developing the study;
12. active autoimmune disease requiring systemic therapy (e.g., use of immunomodulatory agents, corticosteroids, or immunosuppressive agents) was present prior to the initiation of study drug administration, allowing for relevant replacement therapy (e.g., replacement therapy with thyroxine for adrenal or pituitary insufficiency, or physiologic corticosteroids);
13. other malignancies within 5 years prior to the start of study drug administration.
14. a history of previous allogeneic hematopoietic stem cell transplantation or organ transplantation;
15. known hypersensitivity to recombinant humanized anti-HER2 monoclonal antibody-MMAE coupling agent drugs and their components;
16. pregnant or lactating women;
17. estimated to have insufficient patient compliance for participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
12-month disease-free survival (DFS) rate | 12 months after treatment
  Proportion of patients with complete remission confirmed by urine cytology, thoracic-abdominal-pelvic MR, and cystoscopy as a percentage of all patients receiving the full course of medication at 12 months after treatment;

SECONDARY OUTCOMES:
24-month disease-free survival (DFS) rate | 24 months after treatment
  Proportion of patients with complete remission confirmed by urine cytology, thoracic-abdominal-pelvic MR, and cystoscopy as a percentage of all patients receiving the full course of medication at 24 months after treatment;
36-month disease-free survival (DFS) rate | 36 months after treatment
  Proportion of patients with complete remission confirmed by urine cytology, thoracic-abdominal-pelvic MR, and cystoscopy as a percentage of all patients receiving the full course of medication at 36 months after treatment;
disease-free survival (DFS) | From the date of initiation of RC48-based therapy until the date of first documented disease recurrence, progression to muscle-invasive bladder cancer, radical cystectomy, or death from any cause, whichever occurs first, assessed up to 60 months.
overall survival (OS) | From the date of initiation of RC48-based therapy until the date of death from any cause, assessed up to 100 months.

IPD SHARING:
Plan to Share IPD: No